CLINICAL TRIAL: NCT05166824
Title: Clinical Study To Assess The Safety, Parameters And Efficacy For Procedures Using A Radiofrequency Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYN17-RF-CLINIC
Record Dates: First submitted 2021-12-08; First posted 2021-12-22 (Actual); Results first posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Tissue Heating; Coagulation
MeSH Terms: conditions — Thrombosis | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Surgical- abdominoplasty (Experimental): Subjects enrolled in the surgical arm were treated with the device being placed in contact with the skin on the abdomen. The hand piece, number of passes and parameters used for the treatment were determined by the Investigator.
  Interventions: Device: TempSure; Device: Scalpel; Device: Bovie
- Women's Health (Experimental): Subjects enrolled in the women's health were treated with the device in the vaginal and perineal area.
  Interventions: Device: TempSure
- Skin Rejuvenation (Experimental): The hand piece, applicator or tip was placed in contact with the skin. The entire defined treatment area was treated by delivering energy to the skin. The hand piece, number of passes and parameters used for the treatment was determined by the Investigator.
  Interventions: Device: TempSure; Device: Pelleve
- Surgical- blepharoplasty (Experimental): Subjects enrolled in the surgical arm were treated with the device being placed in contact with the skin on the eyelids. The hand piece, number of passes and parameters used for the treatment were determined by the Investigator.
  Interventions: Device: TempSure

INTERVENTIONS:
Device: TempSure — Radiofrequency platform
Device: Scalpel — Cold knife
  Arms: Surgical- abdominoplasty
Device: Bovie — Electrosurgery and electrocautery platform
  Arms: Surgical- abdominoplasty
Device: Pelleve — Radiofrequency platform
  Arms: Skin Rejuvenation

SUMMARY:
The purpose of this study was to develop parameters and assess the safety of the radiofrequency device for a variety of treatments. Treatment results were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female 18 years of age or older.
* Understands and accepts obligation not to receive any other procedures on the treatment area through the length of the study.
* Understands and accepts the obligation and is logistically able to be present for all visits.
* Is willing to comply with all requirements of the study and sign the informed consent document.

Exclusion Criteria:

* Is pregnant or of child bearing potential and not using medically effective birth control or has been pregnant in the last 3 months, currently breast feeding or planning a pregnancy during the course of the study.
* The subject has active or localized systemic infections.
* The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within in the area to be treated 6 months prior to entering this study.
* Any other types of cosmetic treatments in the area to be treated in the past 6 months are cautioned and determined at the discretion of the investigator.
* The subject has a history of keloids.
* The subject has evidence of active systemic or local skin disease that may alter wound healing.
* The subject has scarring or wounds in the treatment area that would interfere with study assessments.
* The subject has a metal implant (such as but not limited to; titanium orbit or metal chin repair) in the face or head that would interfere with study treatment, or subject has an electronic implantable device (such as but not limited to; pacemakers and embedded defibrillators).
* The subject has any condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound study results or may interfere significantly with the subject's participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Civiok, Study Director — Cynosure, Inc.; Sean Doherty, Principal Investigator — Cynosure, Inc.; Raminder Saluja, Principal Investigator — Saluja Cosmetic and Laser Center; Barry DiBernardo, Principal Investigator — New Jersey Plastic Surgery; Edward Jaccoma, Principal Investigator — Excellent Vision; Jeffrey Dell, Principal Investigator — Institute of Female Pelvic Medicine
Locations (5):
- United States (5):
  - Cynosure, Westford, Massachusetts
  - Excellent Vision, Portsmouth, New Hampshire
  - New Jersey Plastic Surgery, Montclair, New Jersey
  - Saluja Cosmetic and Laser Center, Huntersville, North Carolina
  - Institute of Female Pelvic Medicine, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta V, Sharma VK. Skin typing: Fitzpatrick grading and others. Clin Dermatol. 2019 Sep-Oct;37(5):430-436. doi: 10.1016/j.clindermatol.2019.07.010. Epub 2019 Jul 17. PMID 31896400

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Surgical- Abdominoplasty | Women's Health | Skin Rejuvenation | Surgical- Blepharoplasty
Started | 1 | 10 | 68 | 10
Completed | 1 | 10 | 59 | 10
Not Completed | 0 | 0 | 9 | 0

BASELINE CHARACTERISTICS:
Population: Baseline demographic information was not collected for the 1 subject in the surgical-abdominoplasty group.
Groups:
- Surgical- Abdominoplasty: Subjects enrolled in the surgical arm were treated with the device being placed in contact with the abdomen. The hand piece, number of passes and parameters used for the treatment were determined by the Investigator.
  TempSure: Radiofrequency platform
  Scalpel: Cold knife
  Bovie: Electrosurgery and electrocautery platform
- Surgical- Blepharoplasty: Subjects enrolled in the surgical arm were treated with the device being placed in contact with the eye area The hand piece, number of passes and parameters used for the treatment were determined by the Investigator.
  TempSure: Radiofrequency platform
  Scalpel: Cold knife
  Bovie: Electrosurgery and electrocautery platform
- Total: Total of all reporting groups
Arm/Group | Surgical- Abdominoplasty | Women's Health | Skin Rejuvenation | Surgical- Blepharoplasty | Total
Number analyzed (Participants) | 0 | 10 | 68 | 10 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0 | 0 | 0
  Between 18 and 65 years |  | 9 | 64 | 9 | 82
  >=65 years |  | 1 | 4 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The baseline sex of one of the subjects was not collected.
  Participants
    number analyzed (Participants) | 0 | 10 | 67 | 10 | 87
    Female |  | 10 | 61 | 9 | 80
    Male |  | 0 | 6 | 1 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One subject did not have their race/ethnicity collected.
  Participants
    Caucasian: number analyzed (Participants) | 0 | 10 | 67 | 10 | 87
    Caucasian |  | 10 | 60 | 8 | 78
    Asian: number analyzed (Participants) | 0 | 10 | 67 | 10 | 87
    Asian |  | 0 | 1 | 0 | 1
    Hispanic: number analyzed (Participants) | 0 | 10 | 67 | 10 | 87
    Hispanic |  | 0 | 4 | 1 | 5
    African American: number analyzed (Participants) | 0 | 10 | 67 | 10 | 87
    African American |  | 0 | 2 | 0 | 2
    Other (Unspecified): number analyzed (Participants) | 0 | 10 | 67 | 10 | 87
    Other (Unspecified) | 0 | 0 | 0 | 1 | 1
FitzPatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is. The source for this article is cited in the references section. Population: FitzPatrick Skin Type was not taken for the women's health group because it was not applicable. Additionally, 2 subjects did not have their FitzPatrick Skin Type information collected.
  Participants
    number analyzed (Participants) | 0 | 0 | 66 | 10 | 76
    FitzPatrick Skin Type I |  |  | 1 | 0 | 1
    FitzPatrick Skin Type II |  |  | 26 | 1 | 27
    FitzPatrick Skin Type III |  |  | 33 | 9 | 42
    FitzPatrick Skin Type IV |  |  | 4 | 0 | 4
    FitzPatrick Skin Type V |  |  | 0 | 0 | 0
    FitzPatrick Skin Type VI |  |  | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Subject Satisfaction
Description: The subject will be asked their level of satisfaction using a 6-point Likert scale that ranges from "extremely satisfied" to "extremely unsatisfied," with 1 being extremely unsatisfied and 6 being extremely satisfied.
Time Frame: 30 days post final treatment
Population: Some subjects did not complete their 30 day follow up because they withdrew from the study (not because of any serious adverse events), they were lost to follow up, or they could not attend. The subject in the surgical group (abdominoplasty) was not required to complete subject satisfaction, since their participation was for histology purposes only.
Measure: Count of Participants; unit: Participants
Arm/Group | Women's Health | Skin Rejuvenation | Surgical- Blepharoplasty
Number analyzed (Participants) | 10 | 38 | 10
Participants
  Extremely Satisfied | 0 | 6 | 4
  Satisfied | 2 | 14 | 5
  Slightly Satisfied | 4 | 11 | 1
  Slightly Dissatisfied | 2 | 1 | 0
  Dissatisfied | 2 | 4 | 0
  Extremely Dissatisfied | 0 | 2 | 0

2. Primary Outcome: Number of Tissue Samples With Successful Results
Description: This is the number of tissue samples removed by the device (on 1 subject) that has similar histological results to scalpels and cautery devices currently on the market.
Time Frame: Immediately Post Treatment (Same Day)
Population: The other arms of the study did not undergo abdominoplasties or have biopsies taken. Therefore, they do not have results for this outcome measure.
Measure: Number; unit: samples of abdominoplasty
Arm/Group | Surgical- Abdominoplasty
Number analyzed (Participants) | 1
samples of abdominoplasty | 20

ADVERSE EVENTS:
Time Frame: Adverse Events occurring were captured and followed through study completion, an average of 7 months. Subjects were instructed that they may contact the Investigator at any time throughout the course of the study.
Groups:
- Surgical- Blepharoplasty: Subjects enrolled in the surgical arm were treated with the device being placed in contact with the eyelids. The hand piece, number of passes and parameters used for the treatment were determined by the Investigator.
  TempSure: Radiofrequency platform
  Scalpel: Cold knife
  Bovie: Electrosurgery and electrocautery platform
Arm/Group | Surgical- Abdominoplasty | Women's Health | Skin Rejuvenation | Surgical- Blepharoplasty
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/10 | 0/68 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/10 | 0/68 | 0/10
Other Adverse Events (participants affected / at risk) | 0/1 | 0/11 | 39/68 | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Surgical- Abdominoplasty (N=1) | Women's Health (N=11) | Skin Rejuvenation (N=68) | Surgical- Blepharoplasty (N=10)
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 24 | 9
Edema (Skin and subcutaneous tissue disorders) | 0 | 0 | 30 | 9
Skin Burn (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Bleeding (Skin and subcutaneous tissue disorders) | NA | NA | 0 | 6
Itching (Skin and subcutaneous tissue disorders) | NA | NA | 0 | 8
Crusting (Skin and subcutaneous tissue disorders) | NA | NA | 0 | 4
Hardness (Skin and subcutaneous tissue disorders) | NA | NA | 0 | 2
Infection (Infections and infestations) | NA | NA | 0 | 1
Blistering (Skin and subcutaneous tissue disorders) | NA | NA | 0 | 1
Bruisiing (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT05166824/Prot_SAP_000.pdf